CLINICAL TRIAL: NCT02371447
Title: A Phase I/II Open Label Clinical Trial Assessing Safety and Efficacy of Intravesical Instillation of VPM1002BC in Patients With Recurrent Non-muscle Invasive Bladder Cancer After Standard BCG Therapy
Brief Title: VPM1002BC in Recurrent Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 06/14; SNCTP000001181 (Other: SNCTP); 2014-005330-58 (EudraCT Number)
Record Dates: First submitted 2015-02-10; First posted 2015-02-25 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; recurrent non-muscle invasive bladder cancer; VPM1002BC; BCG therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VPM1002BC Induction (Experimental): Phase 1:
  Induction: 6 intravesical instillations of VPM1002BC in 6-12 weeks (dose de-escalation in cohorts of 3-6 patients)
  Phase 2:
  Induction: VPM1002BC at RP2D established in phase I, 6 intravesical instillations in 6-12 weeks (n=39 including patients treated at RPD2 in phase I)
  Maintenance: 3 instillations of VPM1002BC at months 3, 6 and 12
  Interventions: Drug: VPM1002BC

INTERVENTIONS:
Drug: VPM1002BC — Phase 1:
  Induction: 6 intravesical instillations of VPM1002BC in 6-12 weeks (dose de-escalation in cohorts of 3-6 patients)
  Phase 2:
  Induction: VPM1002BC at RP2D established in phase I, 6 intravesical instillations in 6-12 weeks (n=39 including patients treated at RPD2 in phase I)
  Other Names: Mycobacterium bovis BCG∆ureC::Hly+; VPM1002

SUMMARY:
This phase I/II trial will assess the safety and efficacy of intravesical instillation of VPM1002BC in patients with recurrent non-muscle invasive bladder cancer after TURB (transurethral resection of the bladder) and standard BCG therapy. In phase I part of the trial, a 3+3 dose de-escalation design will be applied to determine the recommended phase II dose (RP2D). In phase II part of the trial, a maximum of 39 patients will be treated at RP2D to further assess the preliminary efficacy of VPM1002BC.The efficacy and tolerability of VPM1002BC will be compared to results previously reported for BCG in a similar population. The quality of life will be also investigated as a secondary endpoint. Additional immunology assessments are foreseen as exploratory analyses to investigate the immunogenicity of VPM1002BC.

The Phase II of the trial has been opened on 27.07.2016.

DETAILED DESCRIPTION:
Therapy background

For intermediate/high risk NMIBC clinical guidelines recommend as standard therapy complete transurethral resection of the bladder tumor (s) (TURB), followed by immunotherapy with six weekly intravesical instillations of approx. 5x10E8 CFUs of Bacillus Calmette Guérin (BCG) and maintenance BCG therapy for at least one year. In addition to the prevention of recurrences and progression of NMIBC, the use of BCG as a means of initiating anti-tumor immunity has been shown to prolong overall survival as compared to TURB alone. BCG has also been shown superior to intravesical chemotherapy in combination with BCG maintenance.

Worldwide, more than 200,000 patients are treated with BCG annually, 30-50% of which are likely to recur. While NMIBC incidence has increased over the past decades, death rates remain low due to the efficacy of intravesical BCG therapy. Failure to BCG therapy occurs in 40-50% of patients in terms of disease recurrence or progression. Due to the high risk of disease progression and to the lack of predictive markers for the risk of progression, radical cystectomy is the preferred option for patients failing to respond to a first course of standard BCG therapy, according to current guidelines.

However, a second course of BCG is appropriate for non high-grade and even for some high-grade recurrent tumors. Based on retrospective studies, a second induction course may achieve a 30% to 50% response rate in patients with an initial complete response and in patients with persistent carcinoma in situ (CIS) after a first course of BCG induction therapy. Only a few data are available from prospective studies regarding the outcome of a second BCG therapy cycle after BCG failure. Di Lorenzo et al (2010) reported on 40 patients receiving BCG reinduction: 87.5% of patients failed to respond to BCG re-induction at one year; one patient died of systemic disease, 37.5% of the patients had to undergo cystectomy and 40% underwent radiation therapy plus systemic chemotherapy after 1 year. Of note, these were initially patients unwilling or unfit to undergo cystectomy. In this trial, BCG reinduction was prospectively compared to intravesical chemotherapy with gemcitabine. The results indicated a small benefit for gemcitabine in terms of recurrence-free survival but no difference in terms of progression-free survival. The poor outcome in these patients failing to respond to BCG therapy reflects the unmet medical need for improved bladder sparing treatments after BCG or other intravesical treatment failure. We need better treatment options for patients failing to respond to BCG therapy as these patients are at high risk of cancer progression. Ultimately, improved treatment of these high-risk patients will increase bladder preservation rates and as a consequence, improve quality of life and decrease health costs.

Rationale for performing the trial

Despite the proven efficacy of BCG treatment in patients with NMIBC, recurrence-free and progression-free survival are still poor. Oddens and coworkers (2013) reported ~35-45% of patients recurred by 5 years and ~10-13% of patients progressed. Recurrence and progression to muscle invasive disease lead to additional surgical and radio-oncological interventions including transurethral resection of the bladder (TURB), cystectomy, and chemo-radiotherapy. Improvement in recurrence-free and progression-free survival rates in NMIBC, therefore, would lead to less surgery, better quality of life (QoL), and probably better overall survival.

For those patients failing to a first course of standard BCG therapy, current guidelines recommend radical cystectomy. Alternative options for patients include re-treatment with BCG or intravesical chemotherapy (including multimodal therapy). The earlier the BCG failure, the more probable is the failure of a second BCG cycle. Only few data are available regarding outcome of a second cycle of BCG after BCG failure. Rosevear (2011) reported a 66% complete response after BCG +IFN-α therapy after 6 months of therapy and Di Lorenzo (2010) reported an even worse 6-month recurrence-free survival (RFS) of ~62% (3% at 24 months). As such, better treatment options are not only needed for first line therapy but also for patients with recurrence after a first course of standard BCG therapy.

VPM1002BC is a live genetically modified Mycobacterium bovis BCG that was originally developed as a vaccine against tuberculosis.

VPM1002BC has an innovative mode of action with a unique potential of inducing tumor specific immune responses. VPM1002BC should be at least as potent as the currently used BCG strains in evoking immune responses. Moreover, based on preclinical data, a favourable adverse events profile is expected.

Therefore, the pivotal and final goal of this trial is the testing of VPM1002BC as a safe, well tolerated and efficacious treatment for NMIBC.

VPM1002BC will be tested for safety, efficacy, tolerability and immunogenicity in a phase I/II clinical trial, respectively, in patients with tumor recurrence after standard BCG according to EAU guidelines who are unwilling or unfit to undergo cystectomy. Thus, the reasons to choose this study population are based on the fact that this population has the highest need for innovative treatment and further to establish VPM1002BC as a safe and effective immunotherapy against NMIBC.

A phase I/II design was chosen in order to be able to assess safety and preliminary efficacy and tolerability of VPM1002BC. As the patient population qualifying for the trial is rare and the conventional BCG re-treatment has shown poor and very poor results (see above) we decided to use a single arm design and to compare efficacy and tolerability to reported results. Based on these conditions, the calculated sample size of 39-45 patients has resulted in a reasonable number of patients in terms of recruitment feasibility.

To the best of our knowledge VPM1002BC will be the first in man trial with recombinant intravesical bacteria and the first-in-man intra-bladder application of VPM1002BC.

Trial Treatment

VPM1002BC will be administered once per week as intravesical instillations as follows:

Induction:

- 6 instillations at weekly intervals. First instillation has to be done within 14 days after registration and corresponds to day 1 of the trial treatment schedule (= treatment start).

Maintenance:

* 3 instillations at weekly intervals starting at week 13 from day 1
* 3 instillations at weekly intervals starting at week 25 from day 1
* 3 instillations at weekly intervals starting at week 49 from day 1

Measurements and procedures:

Baseline assessments before trial therapy consist of radiological assessments, transurethral biopsy of the prostatic urethra in men (in case of suspected or previous CIS) followed by staged TUR of the prostate (in case of positive transurethral biopsy of the prostatic urethra ), PPD testing, TURB for histological confirmation of NMIBC (urothelial carcinoma) including second TURB for confirmation of tumor-free state except for pure CIS of the bladder, physical examination, ultrasound of bladder, blood testing for safety parameters, HIV, pregnancy test for women with child-bearing potential.

In phase I, induction therapy, for every weekly instillation: blood assessments for safety parameters (before the instillation and on day after the instillation), urine assessments (Nitrite, urine culture), urine cytology by bladder wash before instillation 1, vital signs (before the instillation and on day after the instillation). In addition, for instillations 1 and 6: assessment of excretion of VPM1002BC in blood, urine and sputum. In phase II, induction therapy, for instillations 1, 3 and 6 (before the instillation): blood assessments for safety parameters, urine assessments (Nitrite, urine culture). In addition, for instillation 1: physical examination including vital signs and weight, urine cytology by bladder wash.

During maintenance therapy (in phase I and II), for instillations 1 and 3 (before the instillation): blood assessments for safety parameters, urine assessments (Nitrite, urine culture). In addition, for each first instillation: physical examination and temperature.

At weeks 12, 24, 36, 48: cystoscopy, urine cytology by bladder wash, physical examination.

The following investigations have to be performed at the end of treatment (week 60): PPD testing, physical examination including vital signs and weight, blood assessments for safety parameters, urine assessments (Nitrite, urine cytology by bladder wash, urine culture), cystoscopy/cytology, abdominopelvic contrast enhanced CT scan.

Adverse events will be recorded continuously throughout the trial treatment. Treatment-related adverse events will be followed-up until resolution or stabilization.

Quality of Life will be assessed at baseline, before start of maintenance and at the end of trial treatment.

During the follow-up phase: survival status, recurrence and progression will be reported every 3 months in the first 2 years and thereafter every 6 months until 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of recurrent NMIBC (urothelial carcinoma) including repeat TURB confirming tumor-free state of the bladder (confirmed by TURB and biopsy) For patients with pure CIS of the bladder no repeat TURB is necessary.
* Negative cytology before start of treatment, except for patients with concomitant CIS.
* Planned treatment starts 2-5 weeks after last TURB
* Pathological grading includes reporting according to WHO 1973 and 2004.
* One previous cycle of intravesical BCG (induction phase with at least 5 instillations ± maintenance) not more than 5 years ago for NMIBC.
* Patients have recurrent high-risk NMIBC for progression.

Exclusion Criteria:

* Current or previous ≥ T2 urothelial carcinoma (UC) of the urinary bladder
* Bladder surgery or traumatic catheterization or TURB within 2 weeks prior to the expected start of trial treatment
* Stress urinary incontinence >I°, severe urge or urge urinary incontinence preventing the patient to keep the IMP in the bladder for at least 1 hour. Residual urinary bladder volume after micturition is > 150 ml.
* Active concomitant malignant conditions except low risk prostate cancer qualifying for active surveillance according to PRIAS criteria (http://www.prostatecancer-riskcalculator.com/active-surveillance-and-prias-study), basal cell skin carcinoma and cervical carcinoma in situ. History of malignancy in the last 3 years except previous NMIBC.
* Primary or secondary immunodeficiencies
* Positive HIV test
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressive drugs or other immune modifying drugs within three months before instillation
* Uncontrollable urinary tract infection, macroscopic haematuria, suspicion of bladder perforation, urethral strictures (if interfering with trial procedures)
* Current and past pelvic radiation and brachytherapy
* Active tuberculosis or other ongoing mycobacterial infection.
* History of anaphylaxis or severe allergic reactions, known allergies to any component of the investigational product, BCG intolerance
* Local and severe allergy (e.g. ulceration, systemic reactions) to PPD test
* Acute fever or fever (>38.5˚C) in the last 7 days before registration
* Simultaneous administration of antituberculous agents and antibiotics that cannot be stopped until registration

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Phase 1: Dose limiting toxicity (DLT) of intravesical VPM1002BC instillations in patients with recurrence after standard BCG therapy in non-muscle-invasive bladder cancer. | within 5 weeks
  Adverse events grade 3 and 4 related to the trial treatment
Phase 2: Recurrence-free rate in the bladder | at 60 weeks
  No visual evidence of cancer in the bladder and negative cytology.

SECONDARY OUTCOMES:
Time to recurrence in the bladder (from registration to tumor recurrence in the bladder) | within 60 weeks
Time to recurrence (from registration to recurrence at local, regional or distant site) | within 60 weeks
Time to progression (from registration to progression). | within 60 weeks
  Progression is defined as a recurrence with an increased stage or grade.
Overall survival calculated from registration until death from any cause | from registration until death (within 6 years)
Adverse events assessed according to NCI CTCAE v4.0. | within 60 weeks
  from registration until 12 weeks after last instillation for patients not completing the overall treatment or after week 60 for patients completing the entire maintenance phase.
Quality of Life assessed by questionnaires | within 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cyrill Rentsch, MD, PhD, Study Chair — University Hospital, Basel, Switzerland; Andreas Wicki, MD, PhD, Study Chair — University Hospital, Basel, Switzerland
Locations (16):
- Germany (6):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum der Ruhr-Universität Bochum, Herne
  - Universitätsklinikum Jena, Jena
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz
  - Klinikum Nürnberg - Universitätsklinik der Paracelsus Medizinischen Privatuniversität, Nuremberg
  - Uniklinik Regensburg, Regensburg
- Switzerland (10):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital, Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre hospitalier universitaire vaudois CHUV, Lausanne
  - Fondazione Oncologia Lago Maggiore, Locarno
  - Kantonsspital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rentsch CA, Thalmann GN, Lucca I, Kwiatkowski M, Wirth GJ, Strebel RT, Engeler D, Pedrazzini A, Huttenbrink C, Schultze-Seemann W, Torpai R, Bubendorf L, Wicki A, Roth B, Bosshard P, Puschel H, Boll DT, Hefermehl L, Roghmann F, Gierth M, Ribi K, Schafer S, Hayoz S. A Phase 1/2 Single-arm Clinical Trial of Recombinant Bacillus Calmette-Guerin (BCG) VPM1002BC Immunotherapy in Non-muscle-invasive Bladder Cancer Recurrence After Conventional BCG Therapy: SAKK 06/14. Eur Urol Oncol. 2022 Apr;5(2):195-202. doi: 10.1016/j.euo.2021.12.006. Epub 2022 Jan 7. PMID 35012889